CLINICAL TRIAL: NCT05816239
Title: LUng voluMe reductIoN by DuAl ENergy CT Evaluation (LUMINANCE) Study
Status: Completed | Type: Observational
Sponsor: Sameer Avasarala (Other)
Responsible Party: Sponsor-Investigator, Sameer Avasarala, Assistant Professor of Medicine, Case Western Reserve University School of Medicine, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Other Study IDs: STUDY20221082
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lung Perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients being evaluated for bronchoscopic lung volume reduction (BLVR).
  Interventions: Procedure: Dual Energy CT

INTERVENTIONS:
Procedure: Dual Energy CT — Patient will receive Dual Energy CT

SUMMARY:
The purpose of this research study is to see if a special CT scan (dual-energy CT) provides useful information in patients undergoing bronchsoscopic lung volume reduction (valve placement for emphysema). The investigators will enroll up to 30 participants in this study from University Hospitals Cleveland Medical Center. All of the participants from this study will undergo their valve procedure at University Hospitals Cleveland Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age at the time of written informed consent) with emphysema who have been deemed appropriate candidates for bronchoscopic lung volume reduction

Exclusion Criteria:

* Patients unable to provide consent
* Patients who are pregnant or nursing
* Women of child-bearing age will undergo pregnancy tests based on University Hospital (UH) standard bronchoscopy pre-procedural testing
* Patients unable to undergo a DECT chest (contraindications to a CT chest with intravenous contrast such as a reported or documented allergy to intravenous (IV) contrast or impaired renal function, defined as the following:
* Glomerular filtration rate (GFR) <90 ml/min/1.73 m2 at the time of initial evaluation if patient age is ≤ 59 years
* GFR <85 ml/min/1.73 m2 if patient age is 60-69 years
* GFR <75 ml/min/1.73 m2 if patient age is ≥70 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 30 patients within the University Hospitals Health System
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-05-24 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Change in lung perfusion as measured by duel-energy computed tomography | Baseline, 8 weeks
Change in walk distance as measured by six-minute walk test | Baseline, 8 weeks
Change in FEV1 as measured by pulmonary function test | Baseline, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Avasarala, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No